CLINICAL TRIAL: NCT05817721
Title: PROTon Pump Inhibitors and Stent OCclusion Rate Of Lumen Apposing Metal Stents (PROTOCOL)
Brief Title: PROTon Pump Inhibitors and Stent OCclusion Rate Of Lumen Apposing Metal Stents
Acronym: PROTOCOL
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Collaborators: Technical University of Munich (Other); Ludwig-Maximilians - University of Munich (Other); University Hospital in Halle (Other); University of Leipzig (Other); University Hospital Heidelberg (Other); Landesklinikum Sankt Polten (Other); University Hospital, Aachen (Other); University of Oldenburg (Other); University of Newcastle Upon-Tyne (Other); Szeged University (Other); University of Pecs (Other); Semmelweis University (Other); University of Ulm (Other); University Hospital Olomouc (Other); Brno University Hospital (Other); University Hospital Regensburg (Other); Klinikum Stadt Hanau (Other); University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Christoph Ammer-Herrmenau, Principal Investigator, University Medical Center Goettingen
Other Study IDs: 2023-02441
Record Dates: First submitted 2023-03-30; First posted 2023-04-18 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Acute Pancreatitis
Keywords: acute pancreatitis; lumen apposing metal stents (LAMS); proton pump inhibitors (PPI)
MeSH Terms: conditions — Pancreatitis | interventions — Proton Pump Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- PPI-group: Patients who received a lumen apposing metal stent (LAMS) for drainage of a walled off necroses (WON) upon acute pancreatitis (AP) and were prescribed proton pump inhibitors (PPI) concomitantly
  Interventions: Drug: Proton pump inhibitor; Device: LAMS-implantation
- Non-PPI-group: Patients who received a lumen apposing metal stent (LAMS) for drainage of a walled off necroses (WON) upon acute pancreatitis (AP) and were not prescribed proton pump inhibitors (PPI) concomitantly
  Interventions: Device: LAMS-implantation

INTERVENTIONS:
Drug: Proton pump inhibitor — Patients who received a lumen apposing metal stent (LAMS) for drainage of a walled off necrosis (WON) upon acute pancreatitis will be divided into a PPI/Non-PPI group depending on if they concomitantly were prescribed a PPI or not
  Groups: PPI-group
Device: LAMS-implantation — Patients who received a lumen apposing metal stent (LAMS) for drainage of a walled off necrosis (WON) upon acute pancreatitis

SUMMARY:
The goal of this observational retrospective cohort study in combination with an expert study is to assess the clinical relevance and management of Lumen apposing metal stent (LAMS)-occlusion and LAMS-occlusion-related complications as well as the influence of proton pump inhibitors (PPI) on LAMS-occlusion.

The main questions this study aims to answer are:

* the individual management of LAMS-occlusion and LAMS-occlusion-related complications in the respective centers participating in the study.
* if there is an association between PPI-intake and LAMS-occlusion and endoscopic necrosectomies.

Participants for the retrospective cohort study will be enrolled retrospectively among European centers with expertise in pancreatology. The expert survey will be distributed European-wide to centers with special expertise in pancreatology.

DETAILED DESCRIPTION:
A common complication of acute pancreatitis is the formation of necrosis in 5-10% of all patients, which leads to an increased overall mortality of 28% for infected necroses. Currently, lumen apposing metal stents (LAMS) are widely used to address necrotic masses. LAMS-occlusion is postulated to be a considerable complication. However, the prevalence, clinical impact and management of LAMS-occlusion-related complications remains uncertain. Moreover, the German guidelines for management of acute pancreatitis do not specify whether a concomitant proton pump inhibitor (PPI)-therapy should be discontinued or not. A recent study suggested a lower rate of LAMS-occlusions, but a higher number of required endoscopic necrosectomies upon concomitant PPI-therapy. Thus, current data are conflicting.

The investigators therefore aim to perform an expert survey and a retrospective cohort study to elucidate the clinical importance of LAMS-occlusion-related complications and the effect of PPI-intake on occlusion. First, a survey will be sent to European centers with special expertise in pancreatology. Here, the investigators aim to assess the number of LAMS applied annually, whether the experts consider occlusion a clinically relevant complication, and whether there are standard operating procedures for LAMS-occlusion and PPI-discontinuation. Second, the investigators will perform a retrospective multicenter cohort study to assess patient data for PPI intake, frequency of LAMS-occlusion and other complications using a RedCap database.

Quality assurance and data checks of the data entered will be performed by the study coordinator after the initial data entry of the participating centers. For missing data, for which the RedCap form cannot be filled out, the online forms comprise extra fields for "missing data". The data entered in the RedCap online survey will stem from paper or electronic case report forms depending which of these are used at the respective centers. Source data verification will be performed by the participating centers themselves upon data entry into the online questionnaires.

A standard operating procedure will be handed out to the participating centers which will feature any information about how data should be entered. Here, the minimum number of patients which needs to be entered into the study in order to participate will be addressed. The maximum of patients who can be entered is dependent on the respective centers; in principle all patients who received a LAMS for drainage of a WON in the respective centers can be included. As the investigators perform a retrospective study, there will be no need to account for reporting of adverse events.

Based on a power calculation of a preliminary in-house dataset from the University Hospital Goettingen the investigators aim to include a total number of 639 patients.

For missing, unavailable, non-reported or uninterpretable data, the RedCap survey will comprise extra fields as described above. In these, the participating researcher can state that data is missing. If this information is essential for the primary or secondary endpoints of our study, the data entry can be excluded from further analyses by the data monitoring committee.

For the statistical analyses of the data gathered from the expert survey the investigators will apply a Fisher/Chi2-test to assess the clinical relevance as well as the clinical management of LAMS-occlusion and LAMS-occlusion-related complications. For the retrospective cohort study, a Chi2-test will be used to address correlations between PPI-intake and LAMS-occlusion. To assess the frequency of occlusion-related-complications, risk factors for LAMS-occlusion beyond PPI-intake and differences in clinical management of LAMS-occlusion in the respective centers, logistic regression/LASSO will be applied.

ELIGIBILITY:
Retrospective cohort study:

Inclusion Criteria:

- Patients in which a Lumen apposing metal stent (LAMS) was applied into a walled off necrosis (WON) as a complication of an acute pancreatitis (AP).

Exclusion Criteria:

* Patients in which a LAMS was applied into a pseudocyst instead of a WON.
* Patients in which a LAMS was used to address a postoperative pancreatic fistula (POPF).
* Patients in which concomitant PPI-treatment was not assessed/not documented.

Expert survey:

Inclusion Criteria:

- European experts (gastroenterological interventionalists) with expertise in pancreatology

Exclusion Criteria:

* Centers which apply less than 10 LAMS per year
* Centers with less than two years experience with LAMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gender criteria: male/female/diverse
Study Population: All patients included in the retrospective cohort study will be from private/public non-academic or academic teaching hospitals in Europe.
  All patients above 18 years of age who received a lumen apposing metal stent (LAMS) for drainage of a walled off necrosis (WON) upon acute pancreatitis will be included.
  Moreover, the expert survey will be distributed to European experts (gastroenterological interventionalists) from private/public non-academic or academic teaching hospitals with special expertise in pancreatology.
Sampling Method: Probability Sample
Enrollment: 893 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Retrospective Cohort Study Primary Outcome Measure Number 1: Association between frequency of LAMS-occlusion and concomitant PPI-intake | Until LAMS-removal, an average of 4 weeks after implantation
  All patients who received a LAMS from the time-point since LAMS have been used at the respective centers will be included. In all patients who received LAMS, their medical records will be checked if a PPI was taken or not. Next, it will be assessed how many patients who took PPIs (PPI-group) had a LAMS-occlusion in comparison with the patients who did not take a PPI (Non-PPI-group). To associate the PPI intake/no PPI intake with LAMS occlusion, we will fit a multiple logistic mixed-effects model including factors potentially affecting the LAMS occlusion rate. As random effects we will include the record identification number and the years of LAMS placement as a surrogate for experience with LAMS.
Retrospective Cohort Study Primary Outcome Measure Number 2: Association between frequency of endoscopic necrosectomy and concomitant PPI-intake | Until LAMS-removal, an average of 4 weeks after implantation
  All patients who received a LAMS from the time-point since LAMS have been used at the respective centers will be included. In all patients who received LAMS, their medical records will be checked if a PPI was taken or not. Next, it will be assessed how many necrosectomy sessions were performed in patients who took PPIs (PPI-group) in comparison with the patients who did not take a PPI (Non-PPI-group). To associate the PPI intake/no PPI intake with the number of endoscopic necrosectomy sessions, we will perform a multiple negative binomial mixed-effects model taking into account counfounders such as the year in which a LAMS was placed.
Expert Survey Primary Outcome Measure Number 1: Assessment of the clinical relevance of LAMS-occlusion and LAMS-occlusion-related complications | Until LAMS-removal, an average of 4 weeks after implantation
  The expert will be asked if he had experiences with complications after total/partial LAMS-occlusion (yes/no). Moreover, the expert will be asked if he would consider these as frequent complications (yes/no). Next, the expert will be asked how frequent he would consider complications after total/partial LAMS-occlusion to occur (scale 0-20%). Finally, the expert will be asked which complications he had witnessed after total/partial LAMS-occlusion (progression of the pancreatic collection, infection of the WON, sepsis, other).
Expert Survey Primary Outcome Measure Number 2: Assessment of the clinical management of LAMS-occlusion in the respective participating centers | Until LAMS-removal, an average of 4 weeks after implantation
  Two clinical cases will be presented. The first case will be suggestive for a total LAMS occlusion with infection/sepsis as a complication consecutive to the stent-occlusion. The second case will be suggestive for a partial LAMS occlusion with no apparent complication. For each case, the expert will be asked if he would consider this a complication (yes/no). Moreover, it will be asked if the expert would remove the LAMS (yes/no), if he would place pigtails over the ostium afterwards (yes/no) and if not what he would do otherwise (endoscopic necrosectomy, place pigtail through the LAMS, disrupted pancreatic duct evaluation via endoscopic retrograde cholangiopancreatography/magnet resonance cholangiopancreatography (ERCP/MRCP), endoscopic papillotomy, other).

SECONDARY OUTCOMES:
Retrospective Cohort Study Secondary Outcome Number 1: Strength of association between PPI intake and the incidence of GI bleeding rates. | Until LAMS-removal, an average of 4 weeks after implantation
  The first secondary aim of this study is to assess the strength of an association between PPI intake and the incidence of GI bleeding rates by performing logistic regression with Firth's correction.
Retrospective Cohort Study Secondary Outcome Number 2: Strength of association between PPI intake and incidence of WON progression on cross sectional imaging. | Until LAMS-removal, an average of 4 weeks after implantation
  The second secondary aim of this study is to assess the strength of an association between PPI intake and the incidence of WON progression on cross sectional imaging by performing logistic regression with Firth's correction.
Retrospective Cohort Study Secondary Outcome Number 3: Strength of association between PPI intake and incidence of superinfection of the WON | Until LAMS-removal, an average of 4 weeks after implantation
  The third secondary aim of this study is to assess the strength of an association between PPI intake and the incidence of superinfection of the WON by performing logistic regression with Firth's correction.
Retrospective Cohort Study Secondary Outcome Number 4: Strength of association between PPI intake and incidence of sepsis events. | Until LAMS-removal, an average of 4 weeks after implantation
  The fourth secondary aim of this study is to assess the strength of an association between PPI intake the incidence of sepsis events by performing logistic regression with Firth's correction.
Retrospective Cohort Study Secondary Outcome Number 5: Strength of association between PPI intake and length of hospital stay (days). | Until LAMS-removal, an average of 4 weeks after implantation
  The fifth secondary aim of this study is to assess the strength of an association between PPI intake and the length of hospital stay (days) by performing logistic regression with Firth's correction.
Expert Survey Secondary Outcome Number 1: To assess if a standard operating procedure (SOP) for follow-up-examinations regarding stent occlusion after LAMS-implantation exists in the respective centers. | Until LAMS-removal, an average of 4 weeks after implantation
  The expert will basked if a SOP for apparative follow-up-examinations after LAMS application exists at their center (yes/no/unknown). Moreover, it will be asked how many follow up examinations are performed (1, 2, 3 or more), at which time-points (<3 days, within 1 week, 2,3,4,5-8 weeks) and how (CT, MRI, gastroscopy, endoscopic ultrasound, abdominal ultrasound) these are performed. Additionally, it will be asked when the LAMS would be removed normally (≤4weeks, 5-8 weeks, ≥9 weeks after implantation). Moreover, it will be asked which procedure is normally followed after LAMS removal (change LAMS to pigtails, just remove the LAMS, other).
Expert Survey Secondary Outcome Number 2: To assess whether the respective clinical center has a SOP regarding LAMS and concomitant PPI-intake. | Until LAMS-removal, an average of 4 weeks after implantation
  The expert will be asked, if proton pump inhibitors are continued/discontinued upon LAMS-application at his/her center (should be discontinued, should be continued with the same dosage, should be continued with another dosage, currently no standard procedure). If the PPI should be continued in another dosage, it will be asked whether it should be continued in half the standard dose, standard dose, double standard dose or more than standard dose. Moreover, it will be asked if any specific PPI should be discontinued and if yes which of the following (Omeprazole, Esomeprazole, Pantoprazole, Lansoprazole, Rabeprazole).
Expert Survey Secondary Outcome Number 3: To assess the experts definition of the term "LAMS-occlusion" in general, as well as the term "partial LAMS occlusion". | Until LAMS-removal, an average of 4 weeks after implantation
  The expert will be asked which of the following potential causes of LAMS occlusion he/she would include in a universal valid definition for reasons of LAMS-occlusion: tissue ingrowth, tissue overgrowth, food impaction, impaction with liquid necrotic debris, impaction with solid necrotic debris, blood clot formation, stent migration, stent kinking, stent compression, stent fracture, other. Moreover, the expert will be asked how he/she would define partial LAMS-occlusion: An occlusion which is still passable with the endoscope; An occlusion in which you can still see through the LAMS with the optics of the endoscope; An occlusion with liquid parts, other.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Hamm, Principal Investigator — Department of Gastroenterology, University Hopsital Goettingen; Christoph Ammer-Herrmenau, MD, Principal Investigator — Department of Gastroenterology, University Hopsital Goettingen; Volker Ellenrieder, Professor, Study Chair — Department of Gastroenterology, University Hopsital Goettingen
Locations (1):
- University Medical Center Goettingen, Goettigen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Collaborators of this study that recruited patients in the PROTOCOL trial may claim access to the final dataset to perform post-hoc studies; these proposals will be reviewed and granted by the steering committee.

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Werge M, Novovic S, Schmidt PN, Gluud LL. Infection increases mortality in necrotizing pancreatitis: A systematic review and meta-analysis. Pancreatology. 2016 Sep-Oct;16(5):698-707. doi: 10.1016/j.pan.2016.07.004. Epub 2016 Jul 9. PMID 27449605
- [Background] Yasuda I, Takahashi K. Endoscopic management of walled-off pancreatic necrosis. Dig Endosc. 2021 Mar;33(3):335-341. doi: 10.1111/den.13699. Epub 2020 Jun 7. PMID 32306430
- [Background] Chandrasekhara V, Barthet M, Deviere J, Bazerbachi F, Lakhtakia S, Easler JJ, Peetermans JA, McMullen E, Gjata O, Gourlay ML, Abu Dayyeh BK. Safety and efficacy of lumen-apposing metal stents versus plastic stents to treat walled-off pancreatic necrosis: systematic review and meta-analysis. Endosc Int Open. 2020 Nov;8(11):E1639-E1653. doi: 10.1055/a-1243-0092. Epub 2020 Oct 22. PMID 33140020
- [Background] Scarpignato C, Gatta L, Zullo A, Blandizzi C; SIF-AIGO-FIMMG Group; Italian Society of Pharmacology, the Italian Association of Hospital Gastroenterologists, and the Italian Federation of General Practitioners. Effective and safe proton pump inhibitor therapy in acid-related diseases - A position paper addressing benefits and potential harms of acid suppression. BMC Med. 2016 Nov 9;14(1):179. doi: 10.1186/s12916-016-0718-z. PMID 27825371
- [Background] Lorenz P, Lynen Jansen P, Beyer G, Hoffmeister A, Lerch MM, Mayerle J. S3-Leitlinie Pankreatitis - Leitlinienreport der Deutschen Gesellschaft fur Gastroenterologie, Verdauungs- und Stoffwechselkrankheiten (DGVS) - September 2021 - AWMF Registernummer 021-003. Z Gastroenterol. 2022 Mar;60(3):e236-e247. doi: 10.1055/a-1713-4244. Epub 2022 Mar 9. No abstract available. German. PMID 35263780
- [Background] Murata A, Ohtani M, Muramatsu K, Matsuda S. Effects of proton pump inhibitor on outcomes of patients with severe acute pancreatitis based on a national administrative database. Pancreatology. 2015 Sep-Oct;15(5):491-496. doi: 10.1016/j.pan.2015.07.006. Epub 2015 Aug 8. PMID 26296720
- [Background] Yoo JH, Kwon CI, Yoo KH, Yoon H, Kim WH, Ko KH, Hong SP, Park PW. [Effect of proton pump inhibitor in patients with acute pancreatitis - pilot study]. Korean J Gastroenterol. 2012 Dec;60(6):362-7. doi: 10.4166/kjg.2012.60.6.362. Korean. PMID 23242019
- [Background] Powers PC, Siddiqui A, Sharaiha RZ, Yang G, Dawod E, Novikov AA, Javia A, Edirisuriya C, Noor A, Mumtaz T, Iqbal U, Loren DE, Kowalski TE, Cosgrove N, Alicea Y, Tyberg A, Andalib I, Kahaleh M, Adler DG. Discontinuation of proton pump inhibitor use reduces the number of endoscopic procedures required for resolution of walled-off pancreatic necrosis. Endosc Ultrasound. 2019 May-Jun;8(3):194-198. doi: 10.4103/eus.eus_59_18. PMID 30719997
- [Background] Martins de Oliveira R, Antunes E, Pedrazzoli J Jr, Gambero A. The inhibitory effects of H+ K+ ATPase inhibitors on human neutrophils in vitro: restoration by a K+ ionophore. Inflamm Res. 2007 Mar;56(3):105-11. doi: 10.1007/s00011-006-6127-6. PMID 17406807
- [Background] Handa O, Yoshida N, Fujita N, Tanaka Y, Ueda M, Takagi T, Kokura S, Naito Y, Okanoue T, Yoshikawa T. Molecular mechanisms involved in anti-inflammatory effects of proton pump inhibitors. Inflamm Res. 2006 Nov;55(11):476-80. doi: 10.1007/s00011-006-6056-4. PMID 17122965
- [Background] Hackert T, Tudor S, Felix K, Dovshanskiy D, Hartwig W, Simon WA, Werner J. Effects of pantoprazole in experimental acute pancreatitis. Life Sci. 2010 Oct 23;87(17-18):551-7. doi: 10.1016/j.lfs.2010.09.008. Epub 2010 Sep 17. PMID 20851132
- [Derived] Hamm J, Busana A, Amanzada A, Arlt A, Asendorf T, Carswell S, Denzer U, Elsing L, Frost F, Guilabert L, Hamesch K, Hollenbach M, Hegyi P, Kleger A, Krivinka J, Kunovsky L, Meinhardt C, Phillip V, Schlosser-Hupf S, Sirtl S, Welsch L, Cardinal von Widdern J, Neesse A, Ammer-Herrmenau C; PROTOCOL working group. Effect of proton pump inhibitors on occlusion of lumen-apposing metal stents and rate of endoscopic necrosectomies: a Europe-wide multicenter cohort study. Endoscopy. 2025 Aug;57(8):829-838. doi: 10.1055/a-2569-7056. Epub 2025 Mar 31. PMID 40164133